CLINICAL TRIAL: NCT02381184
Title: Extended Clomiphene Citrate Regimen Versus Laparoscopic Ovarian Drilling for Ovulation Induction in Clomiphene Citrate-resistant Women With Polycystic Ovary Syndrome
Brief Title: Extended Clomiphene Citrate Regimen in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, principal investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: khalid-walid
Record Dates: First submitted 2015-02-28; First posted 2015-03-06 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene Citrate group (Group A) (Active Comparator): Group A (n =68) assigned to receive100 mg of clomiphene citrate (Clomid®; Hoechst Marion Russel, Cairo, Egypt) daily starting on day 3 of spontaneous or progestin induced cycle for 10 days.
  Interventions: Drug: clomiphene citrate
- laparoscopic ovarian drilling (LOD) Group B (Active Comparator): Group B (n =68) underwent LOD. Laparoscopy was performed under general anesthesia, using three-puncture technique. Each ovary was cauterized perpendicular to its antimesenteric border at four points, each for 4 seconds at 40 W with a mixed current, using a monopolar electrosurgical needle (Karl Storz, ND, Germany). Each puncture was about 4 mm in diameter and 6-8 mm in depth. The ovary was cooled by irrigation with normal saline solution. Any, intraoperative or postoperative complication was reported. The follow-up was started from the next cycle after ovarian drilling up to 6 months
  Interventions: Procedure: laparoscopic ovarian drilling (LOD)

INTERVENTIONS:
Drug: clomiphene citrate — receive100 mg of clomiphene citrate (Clomid®; Hoechst Marion Russel, Cairo, Egypt) daily starting on day 3 of spontaneous or progestin induced cycle for 10 days.
  Other Names: Clomid
  Arms: Clomiphene Citrate group (Group A)
Procedure: laparoscopic ovarian drilling (LOD) — Laparoscopy was performed under general anesthesia, using three-puncture technique
  Arms: laparoscopic ovarian drilling (LOD) Group B

SUMMARY:
One hundred and thirty six anovulatory women with CC-resistant PCOS were scheduled randomly into two equal groups. Group A (n=68); received CC (100 mg/day from cycle day 3 for 10 days) for up to six cycles. Group B (n=68) underwent LOD and followed up for 6 months. The primary outcome was the ovulation rate in each group; secondary outcomes were midcycle endometrial thickness and serum estradiol, midluteal serum progesterone, and the rates of clinical pregnancy and abortion.

DETAILED DESCRIPTION:
This prospective randomized trial included 136 anovulatory women with CC-resistant PCOS among those attending the Gynecology Outpatient Clinics of, Benha University Hospital, and private practice settings, Alkalubia, Egypt from August 2012 to August 2014. The study protocol was approved by the Local Ethics Committee and written informed consents were obtained before the study commenced. Diagnosis of PCOS was based on the Rotterdam criteria (18), whereby diagnosis of PCOS require the presence of two of three criteria after the exclusion of other etiologies, i.e., oligomenorrhea and/or anovulation, clinical and/or biochemical signs of hyperandrogenism, and/or polycystic ovaries on ultrasound. Inclusion criteria: 1- Age: between 18-35 years. 2- Period of infertility > 2 years. 3- Serum level of FSH <10 U/L in the early follicular phase. 4- All women were CC-resistant PCOS, as they failed to ovulate with a dose of CC of 150 mg/day for 5 days per cycle for at least three consecutive cycles. 5- All women had patent Fallopian tubes proved by hysterosalpingography or laparoscopy and their partners satisfied the normal parameters of semen analysis according to the modified WHO criteria (19). Exclusion criteria: 1- Infertility due to causes other than CC- resistant PCOS or due to combined factors. 2- Body mass index (BMI) ≥35 Kg/m². 3- The use of metformin, gonadotropins, hormonal contraception or diet regimen within the last 6 months. 4- Women with congenital adrenal hyperplasia, hyperprolactinaemia or abnormal thyroid function. 5- Hypersensitivity or contraindications to Letrozole or clomiphene treatment. 6- Previous LOD. The study was started two months after last CC treatment cycle to eliminate any post-treatment effect of CC.

At admission, a thorough evaluation of all participants was carried out via history taking and physical examination, which included anthropometric measurements. A baseline transvaginal ultrasound examination was done using 7-10 MHZ probe (Voluson 730 PRO V, GE Healthcare, USA) to measure endometrial thickness and exclude any pelvic pathology before treatment. Basal hormonal assays were performed on day 3 of the spontaneous or progestin induced cycle and included measurement of the serum concentrations of luteinizing hormone (LH), follicle-stimulating hormone (FSH), and testosterone.

Randomization was done according to a computer generated random numerical table into two equal groups. Treatment allocation was concealed by using sequentially numbered opaque sealed envelopes. Envelopes were opened consecutively by a third person (study nurse), who assigned patients to the extended Clomiphene Citrate group (Group A) or LOD group (Group B). Once allocated, the treatment was revealed to both the investigator and the patient. Group A (n =68) assigned to receive100 mg of clomiphene citrate (Clomid®; Hoechst Marion Russel, Cairo, Egypt) daily starting on day 3 of spontaneous or progestin induced cycle for 10 days. Group B (n =68) underwent LOD. Laparoscopy was performed under general anesthesia, using three-puncture technique. Each ovary was cauterized perpendicular to its antimesenteric border at four points, each for 4 seconds at 40 W with a mixed current, using a monopolar electrosurgical needle (Karl Storz, ND, Germany). Each puncture was about 4 mm in diameter and 6-8 mm in depth. The ovary was cooled by irrigation with normal saline solution. Any, intraoperative or postoperative complication was reported. The follow-up was started from the next cycle after ovarian drilling up to 6 months.

Starting from cycle day 9, ultrasound scans were repeated daily to monitor follicle growth (number and mean diameter). Ultrasound examination was done by the same doctor to avoid interobserver variability and he was blinded to the treatment groups. When the optimal follicle size was reached (i.e. mean follicular diameter ≥ 18 mm), HCG 10,000 IU (Epifasi, EPICO, Egypt) was given intramuscular to trigger ovulation. No HCG was given and protected sexual intercourse was advised, if there were ≥ 3 follicles with a diameter ≥16mm to avoid the risk of ovarian hyperstimulation syndrome and multiple gestations. Intrauterine insemination was performed 36 - 40 hours after HCG injection using soft tip catheter.

Serum E2 and the endometrial thickness were measured on the day of HCG administration. The endometrial thickness was measured in a sagittal plane in the fundus of the uterus (point of maximal thickness) from the echogenic interface at the junction of the endometrium and myometrium Ovulation was confirmed when midluteal (day 21of the cycle) serum progesterone was ≥ 5 ng/mL. Serum β-hCG was determined 2 weeks after HCG injection for diagnosis of biochemical pregnancy. Sonographic evidence of an intrauterine gestational sac at 6 weeks gestation was considered an evident of a clinical pregnancy.

Treatment continued for up to six months. Patients were counseled for further lines of treatment if there was no ovulation as confirmed by midluteal serum progesterone level less than 5 ng /ml within 3 months.

The primary outcome was the ovulation rate in each group. Secondary outcomes were the endometrial thickness and serum estradiol (pg/ml), on the day of the hCG injection, midluteal serum progesterone (ng/ml) and the rates of clinical pregnancy and first trimester spontaneous abortion. The ovulation rate was calculated as the percentage of ovulatory cycles per total observed cycles. The cumulative pregnancy rate was defined as the number of pregnant patients to the total number of patients. The abortion rate was defined as the percentage of miscarriage during the first 12 weeks of gestation per total pregnancies, while the biochemical miscarriage was considered if pregnancy loss occurred in any confirmed biochemical pregnancy without ultrasound evidence of intrauterine pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18-35 years
* Period of infertility > 2 years
* Serum level of FSH <10 U/L in the early follicular phase
* All women were CC-resistant PCOS, as they failed to ovulate with a dose of CC of 150 mg/day for 5 days per cycle for at least three consecutive cycles
* All women had patent Fallopian tubes proved by hysterosalpingography or laparoscopy and their partners satisfied the normal parameters of semen analysis according to the modified WHO criteria

Exclusion Criteria:

* Infertility due to causes other than CC- resistant PCOS or due to combined factors
* Body mass index (BMI) ≥35 Kg/m²
* The use of metformin, gonadotropins, hormonal contraception or diet regimen within the last 6 months
* Women with congenital adrenal hyperplasia, hyperprolactinaemia or abnormal thyroid function
* Hypersensitivity or contraindications to Letrozole or clomiphene treatment
* Previous LOD

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
the ovulation rate | midluteal (day 21of the cycle)
  serum progesterone was ≥ 5 ng/mL.

SECONDARY OUTCOMES:
the endometrial thickness | the day of the hCG injection
  Sonographic of endometrial thickness
the rates of clinical pregnancy | 2 weeks after HCG injection
  Serum β-hCG is determined Sonographic evidence of an intrauterine gestational sac at 6 weeks gestation was considered an evident of a clinical pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed morad, Principal Investigator — assistant professor; khalid mohamed, Study Chair — lecturer
Locations (1):
- Benha Faculty of Medicine, Banhā, El Qaluobia, Egypt